CLINICAL TRIAL: NCT02640963
Title: Feasibility and Benefits of Group Based Exercise in Residential Aged Care Adults: a Pilot Study for the GrACE Programme
Brief Title: Feasibility and Benefits of Group Based Exercise in Residential Aged Care Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bond University (Other)
Responsible Party: Principal Investigator, Samantha Fien, Student, Bond University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RO 1823
Record Dates: First submitted 2015-12-15; First posted 2015-12-29 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Geriatric Disorder; Sarcopenia
Keywords: exercise; older adults; physical performance
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention: the GrACE programme (Experimental): The programme included several weight-bearing exercises (using body weight and dumbbells) and a range of seated, non-resisted upper- and lower-body dynamic and reaching movements. While developed for respite care older adults, the GrACE programme was slightly modified for the RAC setting; using reduced range of motion and resistance, and an extended conditioning/familiarisation phase. The conditioning phase lasted for three weeks and focus on the development of correct technique. After concluding the conditioning phase, participants started to use light dumbbells. Participants performed the exercises twice per week for 12 weeks. Training sessions lasted approximately 45 minutes, were separated by at least 48 hours and were delivered by an experienced allied health professional.
  Interventions: Other: Exercise
- Control Group (Placebo Comparator): All subjects assigned to the control group were given the option to engage in other activities that were offered by the facility during the 12-week intervention period. Activities were facility specific, and included Zumba aerobic exercise and walking, however no specific resistance exercises were offered.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — to determine the feasibility of the GrACE (Group Aged Care Exercise) programme in RAC, with the secondary objective of measuring the programme benefits on gait speed, sit to stand and handgrip strength.
  Arms: Intervention: the GrACE programme
Other: Control — to compare with the GrACE (Group Aged Care Exercise) programme in RAC, as well as the secondary objective of measuring the programme benefits on gait speed, sit to stand and handgrip strength against the intervention group
  Arms: Control Group

SUMMARY:
This study is a pilot study (feasibility and acceptability study), which will compare feasibility and efficacy outcomes between a 12-week Exercise Program and control group in RAC residents.

DETAILED DESCRIPTION:
Study Design and Recruitment This study compared the delivery feasibility and outcomes of a 12-week combined resistance and weight bearing exercise programme which the investigators named the GrACE programme. Participant recruitment and assessment occurred over a five-month period.

The RAC was approached about participation via email and telephone follow-up. Potential participants were identified at a meeting with the facility Service Manager. Participants were screened via the inclusion criteria at the meeting with the Service Manager and a Registered Nurse, and written consent was attained prior to participation. Following an explanation of the procedures, purposes, benefits and associated risks of the study, participants had the opportunity to ask questions. A total of 37 older RAC adults provided written informed consent for the study. The exercise group contained 20 participants and the control group 17 participants. Ethical approval to conduct this study was attained from Bond University's Human Ethics Research Committee (RO 1823).

Intervention: the GrACE programme Previous work by our group trialled a successful exercise programme in respite day care that could promise benefits to those in RAC (HenwoodWooding & de Souza 2013). In brief, the GrACE programme included a number of targeted weight-bearing exercises (using body weight and dumbbells) and a range of seated, non-resisted upper- and lower-body dynamic and reaching movements. While developed for respite care older adults, the programme was slightly modified for the RAC setting; initially using reduced range of motion and resistance, and an extended conditioning/familiarisation phase. The conditioning phase lasted for three weeks in which technique was emphasised without using any weights or additional resistance. The focus of this technique of the conditioning phase was to develop the correct technique and minimise the potential for any delayed onset muscle soreness or adverse effects. After concluding the conditioning phase, participants were able to use light dumbbells (often starting with 0.5kg) increasing to heavier dumbbells (up to 4kg) with their increasing capacity over the course of the programme. Participants performed the exercises twice per week for 12 weeks. Training sessions lasted approximately 45 minutes, were separated by at least 48 hours and were delivered by an allied health professional experienced working with RAC adults.

Control Group All subjects assigned to the control group were given the option to engage in other activities that were offered by the facility during the 12-week intervention period. Activities were facility specific, and included Zumba Gold aerobic exercise and walking, however no specific resistance exercises were offered.

Data Collection Reasons for refusal (non-consent) to participate were recorded (Henwood 2014). All muscle function outcome measures in this study have been previously validated for use with older adults, and their protocols reported elsewhere (Henwood, Wooding & de Souza 2013; Sterke et al. 2012). Assessments were completed one-on-one with each participant. During muscle function measures assessments, participants were encouraged to rest as needed and given verbal support and encouragement to reduce any potential burden to the participant.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years and over,
* Residing in a RAC,
* Able to walk with a walker and/or walking stick or could self-ambulate and,
* Could provide informed consent.

Exclusion Criteria:

* End-stage terminal and/or life expectancy <6-months (ethical reasons),
* Two person transfer or unable to self-ambulate (due to increased falls risk),
* Unable to communicate or follow instructions (personal needs beyond the scope of this project),
* Insufficient cognitive function to provide informed consent and,
* Dangerous behaviours that would endanger the client or research staff.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
recruitment rate | up to 12 weeks
  defined as the number of residents recruited from those invited. Measurement units = number and percentage
measurement (physiological and surveys) completion rate | up to 12 weeks
  defined as the number of participants able to complete each outcome measure at baseline and follow-up. Measurement units = number and percentage
loss-to-follow-up | up to 12 weeks
  defined as participants who withdrew or dropped out and did not consent to a follow up assessment. Measurement units = number and percentage
exercise session adherence | up to 12 weeks
  measured by the number of sessions attended out of the maximum 24 sessions. Measurement units = number and percentage
acceptability | up to 12 weeks
  measured via a programme satisfaction survey completed post-training that assessed the burden of training and testing, as well as how participants felt about the trial. Measurement units = number and percentage
adverse events | up to 12 weeks
  defined as incidents in which harm or damage resulted to a participant and included, but were not limited to, falls and fall-related injuries, musculoskeletal or cardiovascular incidents and problems with medication and medical devices. Measurement units = number and percentage

SECONDARY OUTCOMES:
Gait Speed | change from baseline to 12 weeks
  Gait speed was recorded via the GaitMat II system (Manufacturer is EQInc; Model is GaitMat II), which required participants to walk across a level pressure mat system 3.66 m (11.91 ft.) long (McDonough et al. 2001). Participants completed the trials at their preferred (habitual) walking (gait) speed. The following instructions were given, "Walk towards the end of the room at a pace that is comfortable for you". Participants were allowed to walk in their own footwear. All measures were initiated from a standing start 2 m (6.56 ft.) from the GaitMat II platform as suggested by Kressig and Beauchet (Kressig & Beauchet 2006) to reduce the effect that acceleration may have on gait speed. The average gait speed (m/s) from three attempts was used for data analysis. Participants were allowed as much rest as required between attempts, with rest periods typically being up to 1 minute. Measurement units = metres per second
Handgrip strength | change from baseline to 12 weeks
  Upper body muscle function was measured by isometric handgrip strength and sit-to-stand performance, respectively. When performing the handgrip strength assessments, participants were seated, instructed to keep their elbow at 90° and asked to squeeze a handgrip dynamometer (Sammons Preston Roylan, Bolingbrook, IL) to their maximum ability for a period of up to five seconds (Mathiowetz 2002). Three trials were performed with the subject's dominant hand with one-minute rest between trials and the best result used for analysis (Roberts 2011). Measurement units = kilograms
Sit to stand performance | change from baseline to 12 weeks
  In the sit-to-stand measure, participants sat and stood to a full standing position from a chair as many times as possible in 30 seconds whilst keeping their arms crossed against their chest (Millor 2013). Measurement units = repetitions in 30 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Justin Keogh, PhD, Study Chair — Bond University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henwood TR, Keogh JW, Reid N, Jordan W, Senior HE. Erratum to: Assessing sarcopenic prevalence and risk factors in residential aged care: methodology and feasibility. J Cachexia Sarcopenia Muscle. 2014 Sep;5(3):237. doi: 10.1007/s13539-014-0151-0. No abstract available. PMID 24898356
- [Background] McDonough AL, Batavia M, Chen FC, Kwon S, Ziai J. The validity and reliability of the GAITRite system's measurements: A preliminary evaluation. Arch Phys Med Rehabil. 2001 Mar;82(3):419-25. doi: 10.1053/apmr.2001.19778. PMID 11245768
- [Background] Sterke CS, van Beeck EF, Looman CW, Kressig RW, van der Cammen TJ. An electronic walkway can predict short-term fall risk in nursing home residents with dementia. Gait Posture. 2012 May;36(1):95-101. doi: 10.1016/j.gaitpost.2012.01.012. Epub 2012 Mar 3. PMID 22386897
- [Background] Kressig RW, Beauchet O; European GAITRite Network Group. Guidelines for clinical applications of spatio-temporal gait analysis in older adults. Aging Clin Exp Res. 2006 Apr;18(2):174-6. doi: 10.1007/BF03327437. PMID 16702791
- [Background] Mathiowetz V. Comparison of Rolyan and Jamar dynamometers for measuring grip strength. Occup Ther Int. 2002;9(3):201-9. doi: 10.1002/oti.165. PMID 12374997
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] Millor N, Lecumberri P, Gomez M, Martinez-Ramirez A, Izquierdo M. An evaluation of the 30-s chair stand test in older adults: frailty detection based on kinematic parameters from a single inertial unit. J Neuroeng Rehabil. 2013 Aug 1;10:86. doi: 10.1186/1743-0003-10-86. PMID 24059755
- [Background] Henwood T, Wooding A, and de Souza D. 2013. Centre-based exercise delivery: feasability of a staff-delivered program and the benefits for low-functioning older adults accessing respite day care. Activities, Adaptations & Ageing 73:224-238.